CLINICAL TRIAL: NCT06547034
Title: VisR Ultrasound for Noninvasively Interrogating Stromal Collagen Organization in Women as a Breast Cancer Biomarker: Evaluation of Surface Compression in Control Subjects
Brief Title: VisR for Noninvasively Interrogating Stromal Collagen Organization as a Breast Cancer Biomarker: Evaluation of Compression in Control Subjects
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: LCCC2411; 5R01CA281150-02 (NIH)
Record Dates: First submitted 2024-08-01; First posted 2024-08-09 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Breast Cancer
Keywords: Screening
MeSH Terms: conditions — Breast Neoplasms | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Ages 30-45: Women ages 30-45 who have received a mammogram in the past year with negative results and have no history of breast disease.
  Interventions: Device: Ultrasound
- Ages 46-90: Women ages 46-90 who have received a mammogram in the past year with negative results and have no history of breast disease.
  Interventions: Device: Ultrasound

INTERVENTIONS:
Device: Ultrasound — Breast Ultrasound

SUMMARY:
Purpose: The purpose of this study is to evaluate in vivo the diagnostic relevance of ultrasound-derived metrics for elasticity, viscosity, and anisotropy. To this end, we will investigate the effect of applied compression during imaging on elasticity, viscosity, and anisotropy measurements.

Participants: Twenty women with negative mammograms and no history of breast disease will be recruited. The subjects will be split into two cohorts of ten each, the first cohort aged 30-45 and the second cohort aged 46-90. Subjects will be recruited from the Breast Imaging Division of UNC Hospitals.

Procedures (methods): In this exploratory clinical study, the investigators will attempt to demonstrate that ARFI, VisR, and DDAI ultrasound measurements of elasticity, viscosity, and anisotropy in healthy breast tissue vary based on applied pre-compression. This unblinded, open-label study will be conducted in 20 women with negative mammogram results and no history of breast disease.

DETAILED DESCRIPTION:
The primary objective of breast cancer screening is to identify early stage cancer, or precancerous lesions, at a time before symptoms emerge and when treatment is likely to result in a cure. Screening is beneficial when it averts progression of disease to metastasis and/or death, but adverse effects to patients (and unnecessary medical expense) may result downstream from false positives and indiscrimination of masses that will not respond to treatment. The sensitivity of digital mammography, the current screening standard in the US, has been reported in the range of 0.40 to 0.85, with a positive predictive value of 0.31. Sensitivity is increased by augmenting mammography with MRI and B-Mode ultrasound, but false positive rates may also increase. There exists a vital need for a screening technology that exhibits high sensitivity and specificity for cancer detection with early identification of unresponsive masses.

This urgent need could be met by exploiting new imaging biomarkers. Specifically, the mechanical properties of breast tissue have been used for cancer detection, with both elasticity and viscosity demonstrated for discriminating malignant from benign lesions. Further, tissue anisotropy has been shown to correlate with core biopsy result and tumor grade, with large cancers significantly more anisotropic than small cancers. Importantly, while both MRI and ultrasound can be used to measure these biomarkers, ultrasound's cost effectiveness and ease of implementation render it an efficient platform to pursue.

The long-term goal of this research program is to develop a new ultrasound-based breast-screening tool to augment mammography. As a critical first step toward achieving this goal, the primary objective of the proposed research is to evaluate in vivo the replicability of ultrasound-derived metrics for stiffness, elasticity, viscosity, and anisotropy. These biomarkers will be measured using novel, noninvasive ultrasound technologies under development in Dr. Gallippi's laboratory: 1) Acoustic Radiation Force Impulse (ARFI) ultrasound for interrogating tissue stiffness, 2) Viscoelastic Response (VisR) ultrasound for assessing tissue elasticity and viscosity, and 3) Dynamic Displacement Anisotropy Imaging (DDAI) for measuring tissue anisotropy. These technologies have been demonstrated previously for delineating atherosclerosis, muscular dystrophy, and renal dysfunction.

The investigators hypothesize that ultrasound-derived stiffness, elasticity, viscosity, and anisotropy measurements will vary based on applied compression from the sonographer. This is because applying compression to tissue alters its organization, typically reflected by increased stiffness and viscosity and changes in mechanical anisotropy. To test this hypothesis, they will pursue the following specific aim:

Aim #1: Quantify the change in ultrasound-derived stiffness, elasticity, viscosity, and anisotropy measurements from applied pre-compression. ARFI, VisR, and DDAI imaging will be performed on breast stromal tissue in 20 women with negative mammograms and no history of breast disease. Changes in the ultrasound-derived metrics will be evaluated between no applied compression, 10% applied strain, and 25% applied strain. Additionally, magnitude of change in these metrics with applied strain will be compared between two age cohorts (aged 30-45 vs 46-90) and between breast density levels (as rated on BIRADS scale).

ELIGIBILITY:
Inclusion Criteria:

* Patients are 30-90 years of age
* Patients have received a negative result from mammogram screening in past year
* Patients have no history of breast disease
* Informed consent obtained and signed

Exclusion Criteria:

* Inability to provide informed consent
* Inability to communicate in English
* Inability to remain motionless for 15 minutes
* Any pathologies of the breast or history of breast disease
* Patients who are pregnant
* Patients who are lactating
* Patients with breast implants
* Patients with implanted cardioverters or pacemakers

Ages: 30 Years to 90 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Two cohorts of patients with negative mammograms and no history of breast disease will be recruited. Both cohorts will have ten women each. The first cohort will be women ages 30-45, and the second cohort will be women ages 46-90.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2024-10-16 (Actual); Primary Completion 2025-02-28 (Actual); Study Completion 2025-02-28 (Actual)

PRIMARY OUTCOMES:
ARFI PD at 0% Strain | Baseline imaging
  Average ARFI Peak Displacement (PD) value across imaging angles with 0% strain applied. Peak Displacement (PD) - Maximum displacement of tissue in the breast after an Acoustic Radiation Force Impulse (ARFI) excitation.
ARFI PD at 10% Strain | Baseline imaging
  Average ARFI Peak Displacement (PD) value across imaging angles with 10% strain applied. Peak Displacement (PD) - Maximum displacement of tissue in the breast after an Acoustic Radiation Force Impulse (ARFI) excitation.
ARFI PD at 25% Strain | Baseline imaging
  Average ARFI Peak Displacement (PD) value across imaging angles with 25% strain applied. Peak Displacement (PD) - Maximum displacement of tissue in the breast after an Acoustic Radiation Force Impulse (ARFI) excitation.
VisR Tau at 0% Strain | Baseline imaging
  Average VisR Tau value across imaging angles with 0% strain applied. Tau - relaxation constant of breast tissue measured using a Viscoelastic Response (VisR) ultrasound imaging sequence.
VisR Tau at 10% Strain | Baseline imaging
  Average VisR Tau value across imaging angles with 10% strain applied. Tau - relaxation constant of breast tissue measured using a Viscoelastic Response (VisR) ultrasound imaging sequence.
VisR Tau at 25% Strain | Baseline imaging
  Average VisR Tau value across imaging angles with 25% strain applied. Tau - relaxation constant of breast tissue measured using a Viscoelastic Response (VisR) ultrasound imaging sequence.
VisR RE at 0% Strain | Baseline imaging
  Average VisR RE value across imaging angles with 0% strain applied. RE - relative elasticity (relative to force applied) of breast tissue measured using a Viscoelastic Response (VisR) ultrasound imaging sequence.
VisR RE at 10% Strain | Baseline imaging
  Average VisR RE value across imaging angles with 10% strain applied. RE - relative elasticity (relative to force applied) of breast tissue measured using a Viscoelastic Response (VisR) ultrasound imaging sequence.
VisR RE at 25% Strain | Baseline imaging
  Average VisR RE value across imaging angles with 25% strain applied. RE - relative elasticity (relative to force applied) of breast tissue measured using a Viscoelastic Response (VisR) ultrasound imaging sequence.
VisR RV at 0% Strain | Baseline imaging
  Average VisR RV value across imaging angles with 0% strain applied. RV - relative viscosity (relative to force applied) of breast tissue measured using a Viscoelastic Response (VisR) ultrasound imaging sequence.
VisR RV at 10% Strain | Baseline imaging
  Average VisR RV value across imaging angles with 10% strain applied. RV - relative viscosity (relative to force applied) of breast tissue measured using a Viscoelastic Response (VisR) ultrasound imaging sequence.
VisR RV at 25% Strain | Baseline imaging
  Average VisR RV value across imaging angles with 25% strain applied. RV - relative viscosity (relative to force applied) of breast tissue measured using a Viscoelastic Response (VisR) ultrasound imaging sequence.
ARFI PD DoA at 0% Strain | Baseline imaging
  Degree of anisotropy (DoA) defined as ratio of maximum to minimum ARFI Peak Displacement (PD) value across imaging angles with 0% strain applied. Peak Displacement (PD) - Maximum displacement of tissue in the breast after an Acoustic Radiation Force Impulse (ARFI) excitation.
ARFI PD DoA at 10% Strain | Baseline imaging
  Degree of anisotropy (DoA) defined as ratio of maximum to minimum ARFI Peak Displacement (PD) value across imaging angles with 10% strain applied. Peak Displacement (PD) - Maximum displacement of tissue in the breast after an Acoustic Radiation Force Impulse (ARFI) excitation.
ARFI PD DoA at 25% Strain | Baseline imaging
  Degree of anisotropy (DoA) defined as ratio of maximum to minimum ARFI Peak Displacement (PD) value across imaging angles with 25% strain applied. Peak Displacement (PD) - Maximum displacement of tissue in the breast after an Acoustic Radiation Force Impulse (ARFI) excitation.
VisR RE DoA at 0% Strain | Baseline imaging
  Degree of anisotropy (DoA) defined as ratio of maximum to minimum VisR RE value across imaging angles with 0% strain applied. RE - relative elasticity (relative to force applied) of breast tissue measured using a Viscoelastic Response (VisR) ultrasound imaging sequence.
VisR RE DoA at 10% Strain | Baseline imaging
  Degree of anisotropy (DoA) defined as ratio of maximum to minimum VisR RE value across imaging angles with 10% strain applied. RE - relative elasticity (relative to force applied) of breast tissue measured using a Viscoelastic Response (VisR) ultrasound imaging sequence.
VisR RE DoA at 25% Strain | Baseline imaging
  Degree of anisotropy (DoA) defined as ratio of maximum to minimum VisR RE value across imaging angles with 25% strain applied. RE - relative elasticity (relative to force applied) of breast tissue measured using a Viscoelastic Response (VisR) ultrasound imaging sequence.
VisR RV DoA at 0% Strain | Baseline imaging
  Degree of anisotropy (DoA) defined as ratio of maximum to minimum VisR RV value across imaging angles with 0% strain applied. RV - relative viscosity (relative to force applied) of breast tissue measured using a Viscoelastic Response (VisR) ultrasound imaging sequence.

CONTACTS AND LOCATIONS:
Overall Officials: Caterina Gallippi, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol
Time Frame: 9 to 36 months following publication
Access Criteria: The investigator who proposes to use the data has approval from an IRB, IEC, or REB, as applicable, and an executed data use/sharing agreement with UNC.